CLINICAL TRIAL: NCT01146665
Title: Pilot Study of a Computer-Based Intervention for Alcohol Misuse in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Norlien Foundation (Other); Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Principal Investigator, Mandi Newton, Assistant Professor, Department of Pediatrics, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00011650
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Consumption
Keywords: alcohol consumption; personalized assessment feedback; youth; emergency department
MeSH Terms: conditions — Alcohol Drinking; Emergencies

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-based PAF (Experimental): Standard medical care followed by computer-based personalized assessment feedback (PAF).
  Interventions: Behavioral: Computer-based PAF
- Computer-based sham (Sham Comparator): Standard medical care followed by a computer-based sham.
  Interventions: Behavioral: Computer-based Sham

INTERVENTIONS:
Behavioral: Computer-based PAF — This intervention includes standard medical care followed by receipt of computer-based Personalized Assessment Feedback (PAF). PAF is a type of brief intervention that targets norm misperceptions, for example summarizing a person's drinking in comparison to the average male or female in the general population. Theoretically, such normative feedback corrects norm misperceptions and motivates drinkers to re-evaluate their consumption patterns.
  Arms: Computer-based PAF
Behavioral: Computer-based Sham — This intervention includes standard medical care followed by receipt of a computer-based sham. The sham is similar in format and duration as the computer-based Personalized Assessment Feedback but will engage youth in nutrition and exercise-related questions.
  Arms: Computer-based sham

SUMMARY:
Alcohol misuse amongst youth is a significant clinical and public health problem. The Emergency Department (ED) is an important setting for the treatment of alcohol-related problems as it is often the first point of contact between youth, their families, and the healthcare system. This pilot study will assess the feasibility and acceptability of a computer-based intervention in the ED for youth with alcohol-related presentations. The investigators research team will: (1) evaluate the methodological and operational processes involved in study recruitment and intervention implementation, (2) determine recruitment and retention rates, and (3) obtain preliminary data on the difference in alcohol consumption at different time points. The clinical and health service implications of this research will be used to plan further investigations designed to improve the standard of ED care among youth aged 12 to 16 with alcohol-related presentations. This research will also help optimize the planning and development of a full-scale randomized controlled clinical trial of a computer-based intervention designed to reduce higher-risk alcohol consumption and alcohol-related health and social problems in this target population.

ELIGIBILITY:
Study Inclusion Criteria:

* Youth aged 12 to 17 years who present to the Emergency Department (ED) with an alcohol-related problem.
* Medically stable

Alcohol involvement will be determined by youth self-report of drinking alcohol prior to event necessitating a visit to the ED and/or a positive Blood Alcohol Content (BAC).

Study Exclusion Criteria:

* Youth who require hospital admission
* Youth whose ED presentation is linked to drugs aside from alcohol
* Youth who report other drug use within the last 24 hours prior to ED presentation
* Youth who do not speak or understand English
* Youth who are currently enrolled in a treatment program for alcohol use
* Youth who are accompanied by a non-guardianship adult but are not considered Mature Minors
* Youth who do not have the capacity to give informed consent as determined by their attending ED physician
* Youth do not have regular access to their own telephone

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Newton, PhD, Principal Investigator — Faculty of Medicine and Dentistry, University of Alberta; Kathryn Dong, MD, Principal Investigator — Faculty of Medicine and Dentistry, University of Alberta
Locations (3):
- Canada (3):
  - Alberta Children's Hospital Emergency Department, Calgary, Alberta
  - Stollery Children's Hospital Emergency Department, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Derived] Newton AS, Dow N, Dong K, Fitzpatrick E, Cameron Wild T, Johnson DW, Ali S, Colman I, Rosychuk RJ; Pediatric Emergency Research Canada. A randomised controlled pilot trial evaluating feasibility and acceptability of a computer-based tool to identify and reduce harmful and hazardous drinking among adolescents with alcohol-related presentations in Canadian pediatric emergency departments. BMJ Open. 2017 Aug 11;7(8):e015423. doi: 10.1136/bmjopen-2016-015423. PMID 28801399

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Care Plus Computer-based PAF: Computer-based Personalized Assessment Feedback: This brief intervention targeted norm misperceptions, for example summarizing a youth's drinking in comparison to same average male or female in the general population. Theoretically, such normative feedback corrects norm misperceptions and motivates drinkers to re-evaluate their consumption patterns.
- Medical Care Plus Computer-based Sham: Computer-based sham: Similar in format and duration as the Personalized Assessment Feedback but engaged youth in nutrition and exercise-related questions.
Period: Overall Study
Arm/Group | Medical Care Plus Computer-based PAF | Medical Care Plus Computer-based Sham
Started | 18 | 26
1-month Post-ED Discharge (Follow-up) | 9 | 12
3-month Post-ED Discharge (Follow-up) | 8 | 10
Completed | 8 | 10
Not Completed | 10 | 16
Not completed — Withdrawal by Subject | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Standard Medical Care Followed by Computer-based PAF: Standard medical care followed by a brief intervention (computer-based personalized assessment feedback) that targeted norm misperceptions, for example summarizing a youth's drinking in comparison to same average male or female in the general population. Theoretically, such normative feedback corrects norm misperceptions and motivates drinkers to re-evaluate their consumption patterns.
- Standard Medical Care Followed by Computer-based Sham: Standard medical care followed by a computer-based sham intervention. The sham was similar in format and duration as the Personalized Assessment Feedback but engaged youth in nutrition and exercise-related questions.
- Total: Total of all reporting groups
Arm/Group | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham | Total
Number analyzed (Participants) | 18 | 26 | 44
Age, Customized [Count of Participants; unit: Participants]
  13 years | 1 | 2 | 3
  14 years | 3 | 9 | 12
  15 years | 7 | 9 | 16
  16 years | 6 | 6 | 12
  17 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 6 | 7 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 18 | 26 | 44
Met AUDIT-C cut-score of 3 for harmful and hazardous drinking [Count of Participants; unit: Participants] — AUDIT-C (Alcohol Use Disorders Identification Test Consumption subscale): 1 item regarding frequency of alcohol consumption, 1 item regarding the amount of alcohol consumption, and 1 item regarding the frequency of binge drinking. Scores are summed and range from 0 to 12 with higher scores reflecting more consumption. A cut-score of 3 is recommended for identifying youth with harmful and hazardous drinking.
  Participants | 15 | 24 | 39
Report of using other substances prior to ED visit [Count of Participants; unit: Participants]
  Marijuana | 3 | 6 | 9
  Marijuana and ecstasy | 1 | 0 | 1
  Over the counter medication | 0 | 1 | 1
  None | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Youth Alcohol Use
Description: AUDIT-C (Alcohol Use Disorders Identification Test Consumption subscale): 1 item regarding frequency of alcohol consumption, 1 item regarding the amount of alcohol consumption, and 1 item regarding the frequency of binge drinking. Scores range from 0 to 12 with higher scores reflecting more consumption. The change in alcohol use report below reflects the change in AUDIT-C scores with negative values indicating a reduction in score and positive values indicating an increase in score.
Time Frame: baseline, 1 and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Medical Care Followed by Computer-based PAF: Standard medical care followed by a brief intervention (personalized assessment feedback) that targeted norm misperceptions, for example summarizing a youth's drinking in comparison to same average male or female in the general population. Theoretically, such normative feedback corrects norm misperceptions and motivates drinkers to re-evaluate their consumption patterns.
Arm/Group | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 18 | 26
units on a scale
  mean difference from 1 month to baseline | -0.44 (1.34) | -0.88 (1.70)
  mean difference from 3 months to baseline | -0.06 (1.21) | -0.96 (1.82)

2. Secondary Outcome: Recruitment Rate
Description: To be calculated following active recruitment (18 months from study start date of patient enrolment). The recruitment rate relates to recruitment into the study, and not recruitment per arm as randomization and allocation occurred after enrolment.
Time Frame: 18 months
Population: The recruitment rate was calculated as the number of enrolled participants (n=44) divided by the number of eligible participants (n=117).
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The recruitment rate relates to recruitment into the study, and not recruitment per arm as randomization and allocation occurred after enrolment.
Arm/Group | All Participants
Number analyzed (Participants) | 117
Participants
  Number recruited | 44
  Number not recruited | 73

3. Secondary Outcome: Retention Rates
Time Frame: 1 and 3 months post-intervention
Population: We were interested in the overall study retention rates at 1- and 3-months post-intervention, and not retention rates per arm, as the purpose of calculating the rates was to assess the feasibility of a follow-up period in a definitive randomized controlled trial.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The retention rate was calculated as the number participants participating in follow-up data collection divided by the total number of study participants.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Participants
  1 month retention | 21
  3 month retention | 18

4. Secondary Outcome: Knowledge of Treatment Allocation
Time Frame: post-intervention (day 1)
Population: Total number of participants analyzed was 44. Each allocation guess by staff/physicians/nurses was analyzed using the number of adolescents allocated to each arm: 18 to intervention; 26 to control.
Measure: Count of Participants; unit: Participants
Arm/Group | Research Staff | ED Physicians | ED Nurses
Number analyzed (Participants) | 44 | 44 | 44
Participants
  Adolescent was allocated to intervention: number analyzed (Participants) | 18 | 18 | 18
  Adolescent was allocated to intervention: Guess: allocated to intervention | 9 | 5 | 4
  Adolescent was allocated to intervention: Guess: allocated to control | 7 | 0 | 6
  Adolescent was allocated to intervention: Guess: I do not know | 2 | 13 | 8
  Adolescent was allocated to control: number analyzed (Participants) | 26 | 26 | 26
  Adolescent was allocated to control: Guess: allocated to intervention | 16 | 7 | 9
  Adolescent was allocated to control: Guess: allocated to control | 9 | 1 | 3
  Adolescent was allocated to control: Guess: I do not know | 1 | 18 | 14

5. Secondary Outcome: PAF Feasibility and Acceptability
Description: The acceptability of the Personalized Assessment Feedback (PAF) intervention will be assessed by youth post-intervention (only youth allocated to the PAF intervention). Measure assessed acceptability (satisfaction with the intervention, perceptions of the helpfulness, credibility of the personalized assessment feedback) and feasibility (time to completion, user friendliness).
Time Frame: youth: post-intervention (day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Care Plus Computer-based PAF
Number analyzed (Participants) | 18
Participants
  I liked the way the computer program looked: Strongly agreed | 1
  I liked the way the computer program looked: Agreed | 11
  I liked the way the computer program looked: Unsure | 1
  I liked the way the computer program looked: Disagreed | 1
  I liked the way the computer program looked: Strongly disagreed | 0
  I liked the way the computer program looked: Unknown/No response | 4
  This computer program was easy to use: Strongly agreed | 2
  This computer program was easy to use: Agreed | 9
  This computer program was easy to use: Unsure | 1
  This computer program was easy to use: Disagreed | 2
  This computer program was easy to use: Strongly disagreed | 0
  This computer program was easy to use: Unknown/No response | 4
  I was able to finish the computer program quickly: Strongly agreed | 3
  I was able to finish the computer program quickly: Agreed | 8
  I was able to finish the computer program quickly: Unsure | 0
  I was able to finish the computer program quickly: Disagreed | 3
  I was able to finish the computer program quickly: Strongly disagreed | 0
  I was able to finish the computer program quickly: Unknown/No response | 4
  The program helped me think about what I do: Strongly agreed | 1
  The program helped me think about what I do: Agreed | 9
  The program helped me think about what I do: Unsure | 0
  The program helped me think about what I do: Disagreed | 3
  The program helped me think about what I do: Strongly disagreed | 1
  The program helped me think about what I do: Unknown/No response | 4
  The feedback the program gave me was believable: Strongly agreed | 2
  The feedback the program gave me was believable: Agreed | 6
  The feedback the program gave me was believable: Unsure | 3
  The feedback the program gave me was believable: Disagreed | 3
  The feedback the program gave me was believable: Strongly disagreed | 0
  The feedback the program gave me was believable: Unknown/No response | 4

6. Secondary Outcome: Change in Health Care System Utilization by Youth
Description: The Child and Adolescent Services Assessment (CASA) is a self-report instrument designed to assess the use of community- and hospital-based health and social services. We focused each question so that we collected service use for an alcohol use problem.
Time Frame: Baseline
Population: Due to the large amount of missing data (at 1-month [52.3%] and 3-months [59.0%] post-intervention) we did not assess change in utilization from baseline to 1- and 3-months post-intervention (pre-specified secondary outcome) as the results would be prone to bias.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 44 | 18 | 26
Participants
  Hospital: Used (ever) | 3 | 2 | 1
  Hospital: Used in last 3 months | 0 | 0 | 0
  Hospital: Never used | 39 | 15 | 24
  Hospital: Missing | 2 | 1 | 1
  Psychiatrist/Psychologist/SW: Used (ever) | 6 | 3 | 3
  Psychiatrist/Psychologist/SW: Used in last 3 months | 5 | 3 | 2
  Psychiatrist/Psychologist/SW: Never used | 30 | 11 | 19
  Psychiatrist/Psychologist/SW: Missing | 3 | 1 | 2
  Clinic: Used (ever) | 4 | 3 | 1
  Clinic: Used in last 3 months | 1 | 0 | 1
  Clinic: Never used | 37 | 14 | 23
  Clinic: Missing | 2 | 1 | 1
  Crisis service: Used (ever) | 3 | 2 | 1
  Crisis service: Used in last 3 months | 1 | 1 | 0
  Crisis service: Never used | 38 | 14 | 24
  Crisis service: Missing | 2 | 1 | 1
  General physician (GP): Used (ever) | 7 | 6 | 1
  General physician (GP): Used in last 3 months | 2 | 0 | 2
  General physician (GP): Never used | 33 | 11 | 22
  General physician (GP): Missing | 2 | 1 | 1
  School-based service: Used (ever) | 5 | 1 | 4
  School-based service: Used in last 3 months | 4 | 1 | 3
  School-based service: Never used | 33 | 15 | 18
  School-based service: Missing | 2 | 1 | 1
  Family/Friends: Used (ever) | 5 | 3 | 2
  Family/Friends: Used in last 3 months | 8 | 3 | 5
  Family/Friends: Never used | 29 | 11 | 18
  Family/Friends: Missing | 2 | 1 | 1
  Hotline: Used (ever) | 1 | 0 | 1
  Hotline: Used in last 3 months | 1 | 0 | 1
  Hotline: Never used | 40 | 17 | 23
  Hotline: Missing | 2 | 1 | 1
  Self-help: Used (ever) | 0 | 0 | 0
  Self-help: Used in last 3 months | 1 | 1 | 0
  Self-help: Never used | 40 | 16 | 24
  Self-help: Missing | 3 | 1 | 2
  Internet: Used (ever) | 0 | 0 | 0
  Internet: Used in last 3 months | 1 | 1 | 0
  Internet: Never used | 40 | 16 | 24
  Internet: Missing | 3 | 1 | 2

7. Secondary Outcome: Receptivity to Receiving Services: Seeking Help/Treatment
Description: As part of CASA measure (secondary outcome measure to measure health and social services utilization) adolescents were asked two additional questions on receptivity to receiving services. The data below reflects the first question: On a scale of 1-5, where 1 is it's definitely a bad idea and 5 it's definitely a good idea, do you think that if someone you knew had an alcohol use problem they should get help or seek treatment?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 44 | 18 | 26
Participants
  Definitely bad idea | 1 | 0 | 1
  Bad idea | 1 | 1 | 0
  Neutral | 3 | 1 | 2
  Good idea | 10 | 4 | 6
  Definitely good idea | 25 | 10 | 15
  Missing response | 4 | 2 | 2

8. Secondary Outcome: Perceived Barriers to Services
Description: As part of CASA measure (secondary outcome measure to measure health and social services utilization) adolescents answered 8 additional questions on perceived barriers to services: 1) Do you have any feelings such as dislike, distrust or fear about talking with doctors, counselors or other professionals? 2) Do you have any feelings about what other people would think if you sought help? 3) Do you find there is a lack of information that affected health services sought? 4) Do you have any concerns about the amount of time it takes to get help? 5) Were the health services you sought just not readily available? 6) Did you feel you just didn't want to talk to anyone about such a sensitive problem? 7) Was there a problem with registration, setting up appointments or contacting professionals? 8) Was there a problem getting to where treatment was available?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 44 | 18 | 26
Participants
  Negative feelings about talking: No | 16 | 7 | 9
  Negative feelings about talking: Yes, but didn't affect services sought | 7 | 3 | 4
  Negative feelings about talking: Yes and delayed seeking services | 4 | 3 | 1
  Negative feelings about talking: Yes and stopped from seeking services | 0 | 0 | 0
  Negative feelings about talking: Missing | 17 | 5 | 12
  Feelings about what others would think: No | 18 | 8 | 10
  Feelings about what others would think: Yes, but didn't affect services sought | 5 | 2 | 3
  Feelings about what others would think: Yes and delayed seeking services | 3 | 3 | 0
  Feelings about what others would think: Yes and stopped from seeking services | 1 | 0 | 1
  Feelings about what others would think: Missing | 17 | 5 | 12
  Lack of information that affected services sought: No | 24 | 10 | 14
  Lack of information that affected services sought: Yes, but didn't affect services sought | 2 | 2 | 0
  Lack of information that affected services sought: Yes and delayed seeking services | 0 | 0 | 0
  Lack of information that affected services sought: Yes and stopped from seeking services | 0 | 0 | 0
  Lack of information that affected services sought: Missing | 18 | 6 | 12
  Concerns about time it takes to get help: No | 23 | 12 | 11
  Concerns about time it takes to get help: Yes, but didn't affect services sought | 2 | 1 | 1
  Concerns about time it takes to get help: Yes and delayed seeking services | 2 | 0 | 2
  Concerns about time it takes to get help: Yes and stopped from seeking services | 0 | 0 | 0
  Concerns about time it takes to get help: Missing | 17 | 5 | 12
  Health services were not readily available: No | 22 | 11 | 11
  Health services were not readily available: Yes, but didn't affect services sought | 3 | 1 | 2
  Health services were not readily available: Yes and delayed seeking services | 1 | 1 | 0
  Health services were not readily available: Yes and stopped from seeking services | 1 | 0 | 1
  Health services were not readily available: Missing | 17 | 5 | 12
  Didn't want to talk about sensitive problem: No | 16 | 7 | 9
  Didn't want to talk about sensitive problem: Yes, but didn't affect services sought | 3 | 2 | 1
  Didn't want to talk about sensitive problem: Yes and delayed seeking services | 4 | 3 | 1
  Didn't want to talk about sensitive problem: Yes and stopped from seeking services | 3 | 1 | 2
  Didn't want to talk about sensitive problem: Missing | 18 | 5 | 13
  Problem with setting up appointments or contact: No | 22 | 11 | 11
  Problem with setting up appointments or contact: Yes, but didn't affect services sought | 2 | 2 | 0
  Problem with setting up appointments or contact: Yes and delayed seeking services | 1 | 0 | 1
  Problem with setting up appointments or contact: Yes and stopped from seeking services | 0 | 0 | 0
  Problem with setting up appointments or contact: Missing | 19 | 5 | 14
  Problem with getting to where treatment available: No | 23 | 12 | 11
  Problem with getting to where treatment available: Yes, but didn't affect services sought | 2 | 1 | 1
  Problem with getting to where treatment available: Yes and delayed seeking services | 0 | 0 | 0
  Problem with getting to where treatment available: Yes and stopped from seeking services | 0 | 0 | 0
  Problem with getting to where treatment available: Missing | 19 | 5 | 14

9. Secondary Outcome: Receptivity to Services: Doctors/Counselors Can Help
Description: As part of CASA measure (secondary outcome measure to measure health and social services utilization) adolescents were asked two additional questions on receptivity to receiving services. The data below reflects the second question: On a scale of 1-5, where 1 is it's definitely cannot help and 5 it definitely can help, do you think that doctors or counselors can help with alcohol use problems in general?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 44 | 18 | 26
Participants
  Definitely cannot help | 3 | 1 | 2
  Cannot help | 4 | 3 | 1
  Neutral | 8 | 3 | 5
  Can help | 11 | 4 | 7
  Definitely can help | 14 | 5 | 9
  Missing response | 4 | 2 | 2

10. Secondary Outcome: Change in Health Care System Utilization by Youth
Description: as for outcome 6
Time Frame: 1-month post-intervention
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 44 | 18 | 26
Participants
  Hospital: Used (ever) | 0 | 0 | 0
  Hospital: Used in the last 3 months | 2 | 1 | 1
  Hospital: Never used | 19 | 8 | 11
  Hospital: Missing | 23 | 9 | 14
  Psychiatrist/Psychologist/SW: Used (ever) | 1 | 1 | 0
  Psychiatrist/Psychologist/SW: Used in the last 3 months | 5 | 2 | 3
  Psychiatrist/Psychologist/SW: Never used | 15 | 6 | 9
  Psychiatrist/Psychologist/SW: Missing | 23 | 9 | 14
  Clinic: Used (ever) | 1 | 0 | 1
  Clinic: Used in the last 3 months | 3 | 0 | 3
  Clinic: Never used | 17 | 9 | 8
  Clinic: Missing | 23 | 9 | 14
  Crisis service: Used (ever) | 1 | 0 | 1
  Crisis service: Used in the last 3 months | 1 | 1 | 0
  Crisis service: Never used | 19 | 8 | 11
  Crisis service: Missing | 23 | 9 | 14
  General physician (GP): Used (ever) | 1 | 1 | 0
  General physician (GP): Used in the last 3 months | 1 | 0 | 1
  General physician (GP): Never used | 19 | 8 | 11
  General physician (GP): Missing | 23 | 9 | 14
  School-based service: Used (ever) | 1 | 0 | 1
  School-based service: Used in the last 3 months | 3 | 1 | 2
  School-based service: Never used | 17 | 8 | 9
  School-based service: Missing | 23 | 9 | 14
  Family/Friends: Used (ever) | 5 | 3 | 2
  Family/Friends: Used in the last 3 months | 7 | 3 | 4
  Family/Friends: Never used | 9 | 3 | 6
  Family/Friends: Missing | 23 | 9 | 14
  Hotline: Used (ever) | 0 | 0 | 0
  Hotline: Used in the last 3 months | 0 | 0 | 0
  Hotline: Never used | 20 | 9 | 11
  Hotline: Missing | 24 | 9 | 15
  Self-help: Used (ever) | 1 | 0 | 1
  Self-help: Used in the last 3 months | 3 | 2 | 1
  Self-help: Never used | 17 | 7 | 10
  Self-help: Missing | 23 | 9 | 14
  Internet: Used (ever) | 0 | 0 | 0
  Internet: Used in the last 3 months | 0 | 0 | 0
  Internet: Never used | 21 | 9 | 12
  Internet: Missing | 23 | 9 | 14

11. Secondary Outcome: Change in Health Care System Utilization by Youth
Description: as for outcome 6
Time Frame: 3-months post-intervention
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
Number analyzed (Participants) | 44 | 18 | 26
Participants
  Hospital: Used (ever) | 1 | 1 | 0
  Hospital: Used in last 3 months | 1 | 0 | 1
  Hospital: Never used | 15 | 7 | 8
  Hospital: Missing | 27 | 10 | 17
  Psychiatrist/Psychologist/SW: Used (ever) | 2 | 1 | 1
  Psychiatrist/Psychologist/SW: Used in last 3 months | 4 | 2 | 2
  Psychiatrist/Psychologist/SW: Never used | 11 | 5 | 6
  Psychiatrist/Psychologist/SW: Missing | 27 | 10 | 17
  Clinic: Used (ever) | 0 | 0 | 0
  Clinic: Used in last 3 months | 2 | 0 | 2
  Clinic: Never used | 15 | 8 | 7
  Clinic: Missing | 27 | 10 | 17
  Crisis service: Used (ever) | 0 | 0 | 0
  Crisis service: Used in last 3 months | 2 | 1 | 1
  Crisis service: Never used | 15 | 7 | 8
  Crisis service: Missing | 27 | 10 | 17
  General physician (GP): Used (ever) | 1 | 1 | 0
  General physician (GP): Used in last 3 months | 1 | 1 | 0
  General physician (GP): Never used | 11 | 3 | 8
  General physician (GP): Missing | 31 | 13 | 18
  School-based service: Used (ever) | 1 | 1 | 0
  School-based service: Used in last 3 months | 1 | 0 | 1
  School-based service: Never used | 16 | 7 | 9
  School-based service: Missing | 26 | 10 | 16
  Family/Friends: Used (ever) | 0 | 0 | 0
  Family/Friends: Used in last 3 months | 4 | 1 | 3
  Family/Friends: Never used | 14 | 7 | 7
  Family/Friends: Missing | 26 | 10 | 16
  Hotline: Used (ever) | 0 | 0 | 0
  Hotline: Used in last 3 months | 0 | 0 | 0
  Hotline: Never used | 18 | 8 | 10
  Hotline: Missing | 26 | 10 | 16
  Self-help: Used (ever) | 0 | 0 | 0
  Self-help: Used in last 3 months | 1 | 0 | 1
  Self-help: Never used | 16 | 7 | 9
  Self-help: Missing | 27 | 11 | 16
  Internet: Used (ever) | 0 | 0 | 0
  Internet: Used in last 3 months | 0 | 0 | 0
  Internet: Never used | 17 | 7 | 10
  Internet: Missing | 27 | 11 | 16

ADVERSE EVENTS:
Arm/Group | Standard Medical Care Followed by Computer-based PAF | Standard Medical Care Followed by Computer-based Sham
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/26
Other Adverse Events (participants affected / at risk) | 0/18 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No